CLINICAL TRIAL: NCT00249210
Title: A Multicenter, Randomized Study to Compare the Safety and Efficacy of Oral Levofloxacin With Amoxicillin/Clavulanate Potassium in the Treatment of Acute Sinusitis in Adults
Brief Title: A Study of the Safety and Effectiveness of Levofloxacin Compared With Amoxicillin/Clavulanate Potassium in the Treatment of Adults With Rapid Onset of Severe Inflammation/Infection of the Sinuses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005485
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-02

CONDITIONS: Sinusitis; Maxillary Sinusitis
Keywords: Sinusitis; respiratory tract diseases; nose diseases; respiratory tract infections; paranasal sinus diseases; antibacterial agents; quinolones; levofloxacin
MeSH Terms: conditions — Sinusitis; Maxillary Sinusitis; Respiratory Tract Diseases; Nose Diseases; Respiratory Tract Infections; Paranasal Sinus Diseases | interventions — Levofloxacin

INTERVENTIONS:
Drug: levofloxacin

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of levofloxacin, an antibiotic, compared with amoxicillin/clavulanate potassium in the treatment of adults with rapid onset of severe inflammation/infection of the sinuses.

DETAILED DESCRIPTION:
Levofloxacin is an antibacterial agent used for the treatment of many types of severe infections with rapid onset and brief duration in adults. This is a randomized, open-label, parallel group, multicenter study to determine the safety and effectiveness of levofloxacin (500 mg tablets once daily by mouth for 10 - 14 days) compared with amoxicillin/clavulanate (500 mg/125 mg tablets by mouth every 8 hours for 10 - 14 days) in adults with rapid onset of severe inflammation/infection of the sinuses. The study consists of 4 visits: one visit for screening and enrollment, and three visits to assess the safety and effectiveness of treatment (one telephone contact during Days 3 - 6 of the study [if no significant improvement in symptoms has occurred by that time, a visit is scheduled]; one visit [post-therapy] 2 - 5 days after the last dose of the study drug; and one visit [post-study] 28 - 32 days after the last dose of the study drug). The total duration of patient participation in the study is approximately 6 weeks. The primary measure of effectiveness is assessed by the clinical response rate after the completion of treatment (a reduction in the signs and symptoms, and by stabilization or improvement in x-ray findings). Safety evaluations (incidence of adverse events, physical examination, and laboratory tests) are performed throughout the study. The study hypothesis is that treatment with levofloxacin is at least as effective and as well tolerated as treatment with amoxicillin/clavulanate potassium in adults with rapid onset of severe inflammation/infection of the sinuses. 500 mg tablets of levofloxacin by mouth once daily, or 500 mg/125 mg amoxicillin/clavulanate tablets by mouth every 8 hours. The duration of treatment is 10 - 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rapid onset of severe inflammation/infection of the sinuses, as indicated by: fever, headache, discharge from the nose containing pus, facial pain, or tenderness in the area of the cheek bone
* x-ray at the start of the trial consistent with the diagnosis of severe inflammation/infection of the sinuses
* able to take oral medications

Exclusion Criteria:

* Patients with symptoms of sinusitis that has persisted longer than 4 weeks or who have had more than 2 previous episodes of rapid onset of severe inflammation/infection of the sinuses within 12 months prior to the trial
* previous allergic or serious adverse reaction to similar antibiotics
* specific blood and urine test results indicating kidney problems
* requirement of an antibiotic medication taken internally in addition to the study drug or have taken antibiotic medication within 48 hours prior to the start of the study and have experienced improvement
* seizure disorders or any condition requiring tranquilizers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 1993-08; Study Completion 1994-07 (Actual)

PRIMARY OUTCOMES:
Clinical response rate (a reduction in signs and symptoms, and stabilization/improvement of sinus x-ray results) at post-therapy visit, 2 - 5 days after the last dose of study drug

SECONDARY OUTCOMES:
Incidence of adverse events; change in physical examination, and laboratory tests from the start of the study to after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the safety and effectiveness of levofloxacin compared with amoxicillin/clavulanate potassium in the treatment of adults with rapid onset of severe inflammation/infection of the sinuses — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=654&filename=CR005485_CSR.pdf